CLINICAL TRIAL: NCT06455995
Title: Effect of Time-based Energy Intake Goals on Weight Loss During Obesity Treatment
Brief Title: Daily Eating Patterns for Total Health Study
Acronym: DEPTH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Tennessee, Knoxville (Other)
Responsible Party: Principal Investigator, Hollie Raynor, Executive Associate Dean of Research & Operations, College of Education, Health, and Human Sciences, The University of Tennessee, Knoxville
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UTK IRB-23-07697-XP
Record Dates: First submitted 2024-06-06; First posted 2024-06-13 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Meetings will be 60 minutes and led by an interventionist with training at the M.S.- or Ph.D.-level in nutrition, exercise physiology, or behavioral psychology blinded to study hypotheses. Dependent measures will be assessed by a trained researcher blinded to treatment assignment at 0, 3, 6, and 12 months, unless otherwise indicated. The research assistant (blinded to treatment condition) will review all assessment data for accuracy and completion.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- DEPTH-Standard (Active Comparator): Participants in the Standard Group will receive a reduced-energy, low-fat dietary prescription (1200-1500 kcal/d, < 30% energy from fat), physical activity goals (> 200 min/wk of moderate- to vigorous-intensity physical activity [MVPA]) and a cognitive behavioral intervention. Standard group will receive no guidance on energy intake distribution (standard lifestyle intervention).
  Interventions: Behavioral: DEPTH
- DEPTH-Morning (Experimental): Participants in the Morning Group will receive a reduced-energy, low-fat dietary prescription (1200-1500 kcal/d, < 30% energy from fat), physical activity goals (> 200 min/wk of moderate- to vigorous-intensity physical activity [MVPA]) and a cognitive behavioral intervention. They will also have time-based energy intake goals of 70% of kcal within the first 6 hrs of the eating window and 30% of kcal within the last 6 hrs of the eating window (a morning-loaded energy distribution).
  Interventions: Behavioral: DEPTH; Behavioral: DEPTH-Morning
- DEPTH-Evening (Experimental): Participants in the Evening Group will receive a reduced-energy, low-fat dietary prescription (1200-1500 kcal/d, < 30% energy from fat), physical activity goals (> 200 min/wk of moderate- to vigorous-intensity physical activity [MVPA]) and a cognitive behavioral intervention. They will also have time-based energy intake goals of 30% of kcal within the first 6 hrs of the eating window and 70% of kcal within the last 6 hrs of the eating window (an evening-loaded energy distribution).
  Interventions: Behavioral: DEPTH; Behavioral: DEPTH-Evening

INTERVENTIONS:
Behavioral: DEPTH — All conditions will receive a reduced-energy, low-fat dietary prescription (1200-1500 kcal/d, < 30% energy from fat), physical activity goals (> 200 min/wk of moderate- to vigorous-intensity physical activity [MVPA]) and a cognitive behavioral intervention. To minimize the effect of other eating temporal variables on outcomes, guidance on the eating window length and the number of eating occasions in the day will be consistent across all three conditions. Thus, the three conditions will be instructed to have their first eating occasion < 60 minutes of awakening, and eat their three meals and one snack within a 12-hr eating window.
Behavioral: DEPTH-Morning — Morning will also have time-based energy intake goals of 70% of kcal within the first 6 hrs of the eating window and 30% of kcal within the last 6 hrs of the eating window (a morning-loaded energy distribution).
  Arms: DEPTH-Morning
Behavioral: DEPTH-Evening — Evening will also have time-based energy intake goals of 30% of kcal within the first 6 hrs of the eating window and 70% of kcal within the last 6 hrs of the eating window (an evening-loaded energy distribution).
  Arms: DEPTH-Evening

SUMMARY:
The goal of this randomized controlled trial is to learn how the time of day when calories are eaten affects weight loss in the long-term (12 months). The main aims are to learn:

1. The influence of time-based energy intake goals on longer-term weight loss.
2. The influence of time-based energy intake goals on eating temporal patterns, sleep regularity, and appetite regulation.

Researchers will compare whether goals to eat most of a person's calories in the morning or evening work to treat obesity.

Participants will:

1. Eat a reduced-calorie, low-fat diet (some participants will have goals to eat their calories at certain times of day based on their group)
2. Be physically active at least 200 minutes
3. Receive a cognitive behavioral intervention

DETAILED DESCRIPTION:
This randomized controlled trial investigates the longer-term (12 months) effect of time-based energy intake goals on weight loss. It also explores whether enhanced appetite regulation is a mediator of the relationship and if chronotype moderates the effect. Adults with overweight or obesity are randomly assigned to one of three, 12-month lifestyle interventions: 1) Morning; 2) Evening; or 3) Standard. All conditions receive a reduced-energy, low-fat dietary prescription (1200-1500 kcal/d, < 30% energy from fat), physical activity goals (> 200 min/wk of moderate- to vigorous-intensity physical activity [MVPA]) and a cognitive behavioral intervention. To minimize the effect of other eating temporal variables on outcomes, guidance on the eating window length and the number of eating occasions in the day are consistent across all three conditions. Thus, the three conditions are instructed to have their first eating occasion < 60 minutes of awakening, and eat their three meals and one snack within a 12-hr eating window. Morning group has time-based energy intake goals of 70% of kcal within the first 6 hrs of the eating window and 30% of kcal within the last 6 hrs of the eating window (a morning-loaded energy distribution). Evening group has the opposite time-based energy intake goals (an afternoon/evening-loaded energy distribution). Standard group receives no guidance on energy intake distribution (standard lifestyle intervention). Assessments occur at 0, 3, 6, and 12 months on anthropometrics, diet (24-hr recalls with time-stamped digital images verifying timing of intake, combined with continuous blood glucose monitoring [CGM] to objectively assess for length of the eating window and number of eating occasions), sleep regularity (actigraphy supported by sleep logs collected via ecological momentary assessment [EMA] using smartphones), appetite regulation assessed via EMA using smartphones, chronotype (self-reported midpoint of sleep on work-free days), and MVPA (actigraphy).

The primary aims are to determine:

1. The influence of time-based energy intake goals on longer-term weight loss.
2. The influence of time-based energy intake goals on eating temporal patterns, sleep regularity, and appetite regulation.

The exploratory aims are to consider:

1. If appetite regulation mediates the relationship between time-based energy intake goals and weight loss.
2. The moderating effect of chronotype on weight loss and changes in eating temporal patterns, sleep regularity, and appetite regulation in the three conditions.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 27 and 45 kg/m2.

Exclusion Criteria:

* Report not regularly (>/= 5 days/wk) consuming energy (>/= 100 kcal) prior to 12 pm, and not being able to consume energy every day (>/= 50 kcal) within one hour of awakening.
* Report taking sleep medication or not regularly (>/= 5 nights/wk) getting at least 6 hrs of total sleep.
* Report being a shift workers/alternative shift workers that work outside of 7 am and 7 pm.
* Report being diagnosed with type 1, or type 2 diabetes and taking medication that requires eating to occur at certain time periods.
* Report a heart condition, chest pain during periods of activity or rest, or loss of consciousness on the Physical Activity Readiness Questionnaire (PAR-Q). Individuals reporting joint problems, prescription medication usage, or other medical conditions that could limit exercise will be required to obtain written physician consent to participate.
* Report being unable to walk for 2 blocks (1/4 mile) without stopping.
* Report major psychiatric diseases or organic brain syndromes.
* Report currently participating in a weight loss program and/or taking weight loss or appetite regulation medication or lost >/= 5% of body weight during the past 6 months.
* Report having bariatric surgery for weight loss/planning to have bariatric surgery in the next 12 months.
* Report being pregnant, lactating, < 6 months post-partum or plan to become pregnant (next 12 months).
* Report planning to move outside of the metropolitan area within the time frame of the investigation.
* Do not have daily access to PC with internet or smartphones (needed for self-monitoring).

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 174 (Estimated)
Dates: Start 2024-07-16 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Percent Weight Change | 0, 3, 6, and 12 months
  Percent change in weight (weight change in lbs at follow up / baseline weight in lbs)
Body Mass Index (BMI) | 0, 3, 6, and 12 months
  Change in BMI calculated as weight in kg / height in m2

SECONDARY OUTCOMES:
Dietary intake | 0, 3, 6, and 12 months
  Dietary intake will be assessed by 3 (2 weekdays and 1 weekend day), random, 24-hr dietary phone recalls, using the five-step, multiple-pass method
Sleep | 0, 3, 6, and 12 months
  Hours of daily sleep objectively measured by accelerometry
Appetite regulation | 0, 3, 6, and 12 months
  Time- and semi-random sampling will be initiated via a smartphone tone, prompting participants to complete ratings (i.e. hunger, fullness, temptation to eat, desire to eat, and control over eating), using 100 mm visual analogue scales
Waist circumference | 0, 3, 6, and 12 months
  Change in waist circumference in inches
Moderate- to vigorous-physical activity (MVPA) | 0, 3, 6, and 12 months
  Time in MVPA objectively measured by accelerometry
Chronotype | 0, 3, 6, and 12 months
  An individuals' circadian state (phase relationship between the circadian system of an individual and the zeitgeber cycle) measured via the shortened version of the Munich ChronoType Questionnaire

OTHER OUTCOMES:
Process evaluation: Self-monitoring of diet | Throughout the 12-month intervention
  Achievement of condition specific diet goals (adherence) will be documented (days/wk for overall energy and fat goal [staying with + 5% of each goal]; first eating occasion < 60 minutes of awakening; daily eating window length < 12 hours; four eating occasions per day; and time-based energy intake goals [staying within + 5% of each goal] for Morning and Evening only)
Process evaluation: Self-monitoring of physical activity | Throughout the 12-month intervention
  From physical activity self-monitoring records, number of weeks minutes that MVPA is within + 5% of the goal will be documented.
Process evaluation: Attendance | Throughout the 12-month intervention
  Number of sessions attended will be recorded
Process evaluation: Fidelity | Throughout the 12-month intervention
  All sessions will be audiotaped and the PI will review 33% of these sessions for treatment fidelity

CONTACTS AND LOCATIONS:
Locations (1):
- Healthy Eating and Activity Laboratory, Knoxville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Types and amount of scientific data expected to be generated in the project:
  Demographic, anthropometric, dietary intake, sleep and physical activity from actigraphy, appetite regulation collected via ecological momentary assessment, and chronotype data will be collected from 174 adults with overweight or obesity (described in detail in section c.3. of this application) at four time points (0, 3, 6, and 12 months). Raw data will be transformed by processing software (diet and actigraphy) and will generate 4 data sets (data organized by timepoint), which will be no more than 100 gigabytes. These four data sets will be used for statistical analyses and be placed in the repository. All data will be de-identified prior to receipt by the repository, and individual-level data will be made available for sharing.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available as soon as possible or at the time of associated publication, whichever comes first. Data on Dryad are retained indefinitely.
Access Criteria: Dataset(s) resulting from this research will be shared via the generalist repository Dryad, which provides metadata, persistent identifiers (i.e., DOIs), and long-term access. Dryad is the institutional data repository supported by the University of California and all data is shared under a CC0 waiver, which makes the dataset(s) publicly available. Data will be made available as soon as possible or at the time of associated publication. Dryad datasets are backed up to Merritt, the UC's CoreTrustSeal-certified digital repository, for long-term storage and accessibility. Procedures in place to ensure dataset preservation include storage of data files in multiple geographic locations, regular audits for fixity and authenticity, and succession plans in the event of repository closure.
URL: https://cdlib.org/services/uc3/dryad/

REFERENCES:
- [Background] Yong YN, Henry CJ, Haldar S. Is There a Utility of Chrono-Specific Diets in Improving Cardiometabolic Health? Mol Nutr Food Res. 2022 Sep;66(17):e2200043. doi: 10.1002/mnfr.202200043. Epub 2022 Jul 20. PMID 35856629
- [Background] Salgado-Delgado R, Tapia Osorio A, Saderi N, Escobar C. Disruption of circadian rhythms: a crucial factor in the etiology of depression. Depress Res Treat. 2011;2011:839743. doi: 10.1155/2011/839743. Epub 2011 Aug 8. PMID 21845223
- [Background] Petersen MC, Gallop MR, Flores Ramos S, Zarrinpar A, Broussard JL, Chondronikola M, Chaix A, Klein S. Complex physiology and clinical implications of time-restricted eating. Physiol Rev. 2022 Oct 1;102(4):1991-2034. doi: 10.1152/physrev.00006.2022. Epub 2022 Jul 14. PMID 35834774
- [Background] Wang JB, Patterson RE, Ang A, Emond JA, Shetty N, Arab L. Timing of energy intake during the day is associated with the risk of obesity in adults. J Hum Nutr Diet. 2014 Apr;27 Suppl 2:255-62. doi: 10.1111/jhn.12141. Epub 2013 Jun 27. PMID 23808897
- [Background] Hermenegildo Y, Lopez-Garcia E, Garcia-Esquinas E, Perez-Tasigchana RF, Rodriguez-Artalejo F, Guallar-Castillon P. Distribution of energy intake throughout the day and weight gain: a population-based cohort study in Spain. Br J Nutr. 2016 Jun;115(11):2003-10. doi: 10.1017/S0007114516000891. Epub 2016 Apr 5. PMID 27044416
- [Background] Maukonen M, Kanerva N, Partonen T, Mannisto S. Chronotype and energy intake timing in relation to changes in anthropometrics: a 7-year follow-up study in adults. Chronobiol Int. 2019 Jan;36(1):27-41. doi: 10.1080/07420528.2018.1515772. Epub 2018 Sep 13. PMID 30212231
- [Background] Keim NL, Van Loan MD, Horn WF, Barbieri TF, Mayclin PL. Weight loss is greater with consumption of large morning meals and fat-free mass is preserved with large evening meals in women on a controlled weight reduction regimen. J Nutr. 1997 Jan;127(1):75-82. doi: 10.1093/jn/127.1.75. PMID 9040548
- [Background] Jakubowicz D, Barnea M, Wainstein J, Froy O. High caloric intake at breakfast vs. dinner differentially influences weight loss of overweight and obese women. Obesity (Silver Spring). 2013 Dec;21(12):2504-12. doi: 10.1002/oby.20460. Epub 2013 Jul 2. PMID 23512957
- [Background] Rabinovitz HR, Boaz M, Ganz T, Jakubowicz D, Matas Z, Madar Z, Wainstein J. Big breakfast rich in protein and fat improves glycemic control in type 2 diabetics. Obesity (Silver Spring). 2014 May;22(5):E46-54. doi: 10.1002/oby.20654. Epub 2013 Dec 6. PMID 24311451
- [Background] Lombardo M, Bellia A, Padua E, Annino G, Guglielmi V, D'Adamo M, Iellamo F, Sbraccia P. Morning meal more efficient for fat loss in a 3-month lifestyle intervention. J Am Coll Nutr. 2014;33(3):198-205. doi: 10.1080/07315724.2013.863169. Epub 2014 May 8. PMID 24809437

DOCUMENTS (1):
  • Informed Consent Form (2024-06-11): https://cdn.clinicaltrials.gov/large-docs/95/NCT06455995/ICF_001.pdf